CLINICAL TRIAL: NCT05998603
Title: Pre-sleep Protein Supplementation Does Not Improve Recovery From Load Carriage in British Army Recruits
Brief Title: Pre-sleep Protein Supplementation and Load Carriage Recovery in British Army Recruits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1076/MODREC/20B
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Protein-energy; Imbalance; Muscle Soreness
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High protein intake supplementation (Experimental): A 60g daily dose of whey protein supplementation
  Interventions: Dietary Supplement: High protein intake
- Moderate protein intake supplementation (Experimental): A 20g dose of whey protein supplementation
  Interventions: Dietary Supplement: Moderate protein intake
- Carbohydrate placebo (Placebo Comparator): An isocaloic maltodextrin carbohydrate placebo
  Interventions: Dietary Supplement: Carbohydrate maltodextrin placebo
- Control group, no supplementation (Other): Control group, not taking any supplementation, only completing basic training activities
  Interventions: Other: Control no supplementation

INTERVENTIONS:
Dietary Supplement: High protein intake — The participants received a 60g whey protein bolus each evening prior to sleep pre and post a military load carriage test.
  Arms: High protein intake supplementation
Dietary Supplement: Moderate protein intake — The participants received a 20g whey protein bolus each evening prior to sleep pre and post a military load carriage test.
  Arms: Moderate protein intake supplementation
Dietary Supplement: Carbohydrate maltodextrin placebo — The participants received an isocaloric carbohydrate bolus each evening prior to sleep pre and post a military load carriage test.
  Arms: Carbohydrate placebo
Other: Control no supplementation — Control group, no supplementation, only basic training
  Arms: Control group, no supplementation

SUMMARY:
Load carriage is a common military activity and has been shown to induce acute exercise-induced muscle damage (EIMD) and impair muscle function. Protein supplementation can accelerate muscle recovery by attenuating EIMD and muscle function loss. This study investigated the impact of an additional daily bolus of protein prior to sleep throughout training on acute muscle recovery following a load carriage test in British Army recruits. Muscle function (maximal jump height), perceived muscle soreness and urinary markers of muscle damage were assessed before (PRE), immediately post (POST), 24-hours post (24h-POST) and 40-hours post (40h-POST) a load carriage test.

DETAILED DESCRIPTION:
British Army basic training (BT) is physically demanding with new recruits completing multiple bouts of physical activity each day with limited recovery. Load carriage is one of the most physically demanding BT activities and has been shown to induce acute exercise-induced muscle damage (EIMD) and impair muscle function. Protein supplementation can accelerate muscle recovery by attenuating EIMD and muscle function loss. This study investigated the impact of an additional daily bolus of protein prior to sleep throughout training on acute muscle recovery following a load carriage test in United Kingdom (UK) British Army recruits. A mixed group (men/women) over over 120 new recruits were randomised to dietary control (CON), carbohydrate placebo (PLA), moderate (20g; MOD) or high (60g; HIGH) protein supplementation. Muscle function (maximal jump height), perceived muscle soreness and urinary markers of muscle damage were assessed before (PRE), immediately post (POST), 24-hours post (24h-POST) and 40-hours post (40h-POST) a load carriage test. The underlying aim of this study was to assess whether additional protein intake could attenuate aspects of muscle damage from an acute load carriage test including muscle function, muscle soreness and biomarkers of muscle damage during short term recovery.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled into British Army basic training
* Medically fit to train and complete the load carriage test

Exclusion Criteria:

* Not taking any other nutritional supplement
* Pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in lower body muscle function | 40-hours
  The change in maximal vertical jump height in participants before and after the load carriage test

SECONDARY OUTCOMES:
The change in urinary myoglobin | 40-hours
  The relative change in concentration of urinary myoglobin (ng/ml) in participants before and after the load carriage test
The change in urinary 3-methylhistidine | 40-hours
  The relative change in concentration of urinary 3-methylhistidine (nmol/ml) in participants before and after the load carriage test
The change in perceived muscle soreness | 40-hours
  The relative change in perceived muscle soreness assessed via visual analogue scale. The participants were asked to record their perceived muscle soreness using a 0-10 Likert scale (e.g., 0=no pain, 10=severe pain that limits the ability to move).

CONTACTS AND LOCATIONS:
Overall Officials: Justin D Roberts, PhD, Principal Investigator — Anglia Ruskin University
Locations (1):
- Anglia Ruskin University, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No